CLINICAL TRIAL: NCT01495494
Title: A Multiple Use Tolerability Study of a Breathe Right Nasal Strip Prototype
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B3560692
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Subjects
Keywords: Nasal Strip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marketed nasal strip (Active Comparator): Marketed nasal strip
  Interventions: Device: Marketed Nasal Strip
- Prototype nasal dilator (Experimental): Prototype nasal dilator
  Interventions: Device: Prototype Nasal Dilator

INTERVENTIONS:
Device: Marketed Nasal Strip — Breathe Right Nasal Strips - Clear small/medium strip
  Arms: Marketed nasal strip
Device: Prototype Nasal Dilator — Prototype Nasal Dilator AB2R11
  Arms: Prototype nasal dilator

SUMMARY:
This study evaluated the safety & tolerability of two Breathe Right nasal strip prototypes. Prototypes were produced as an improvement to the currently marketed product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Dermal response score of the application site of the nasal strip | Baseline through 7 days

SECONDARY OUTCOMES:
Subjective questionnaire regarding comfort, overnight adherence, and ease of removal of the strip | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Essex Testing Clinic, Inc, Verona, New Jersey, United States

REFERENCES:
- [Derived] Ward J, Ciesla R, Becker W, Shanga GM. Randomized Trials of Nasal Patency and Dermal Tolerability With External Nasal Dilators in Healthy Volunteers. Allergy Rhinol (Providence). 2018 Oct 5;9:2152656718796740. doi: 10.1177/2152656718796740. eCollection 2018 Jan-Dec. PMID 30305980